CLINICAL TRIAL: NCT00595634
Title: Intramedullary Nailing for Treatment of Unstable InterTrochanteric (INTUIT) Hip Fracture Outcome Study.
Brief Title: INTUIT Hip Fracture Outcome Study
Acronym: INTUIT
Status: Terminated | Type: Observational
Why Stopped: Could not power primary endpoint due to lost to follow-up rate
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 03618-07-A
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Unstable Intertrochanteric Hip Fractures
Keywords: Hip; Fracture; Intertrochanteric; intramedullary
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to characterize patients' course of recovery in the year following the initial surgery for unstable intertrochanteric hip fractures treated with the InterTAN intramedullary hip screw device. This will be done by collecting patient outcome measures of health related quality of life and functional status including return to normal gait. Secondary objectives are to document any adverse events associated with the procedure, and to analyze differences in recovery due to differences in age, gender, co-morbidities, nutrition, residence and ambulation status, and use of mobility aids.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral unstable intertrochanteric hip fracture without other lower extremity fractures.
* Community and household ambulators with or without assistive devices.
* Age 50 years or greater.

Exclusion Criteria:

* Stable intertrochanteric hip fracture.
* Bilateral or two or more lower extremity fractures.
* Non-functional ambulators or non-ambulators.
* Age less than 50 years.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with unilateral unstable intertrochanteric hip fracture (as defined by Hennepin County Medical Center intertrochanteric hip fracture classification system, Kyle et al, 1979) without other lower extremity fractures.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2008-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Mobility function as defined by the Timed Up & Go (TUG) frequency. | Baseline, Post-Operatively at 2 Weeks, 6 Weeks, 3 Months, 6 Months and 12 Months

SECONDARY OUTCOMES:
Lower Extremity Activity Scale | Baseline, Post-Operatively at 2 Weeks, 6 Weeks, 3 Months, 6 Months and 12 Months
EuroQol | Baseline, Post-Operatively at 2 Weeks, 6 Weeks, 3 Months, 6 Months and 12 Months
Visual Analogue Score (VAS) | Baseline, Post-Operatively at 2 Weeks, 6 Weeks, 3 Months, 6 Months and 12 Months
Adverse Event | When necessary

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Brown, M.D., Principal Investigator — TRIA Orthopaedic Center, Park Nicollet Health Services
Locations (5):
- United States (5):
  - Sonoran Orthopaedic Trauma Surgeons, PLLC, Scottsdale, Arizona
  - University of California, Irvine, Orange, California
  - Shrock Orthopedic Research, LLC, Fort Lauderdale, Florida
  - Orthopaedic Center of Vero Beach, Vero Beach, Florida
  - Park Nicollet, Saint Louis Park, Minnesota

REFERENCES:
- See also: TRIA Orthopaedic Center — http://www.tria.com/